CLINICAL TRIAL: NCT00643058
Title: Nitric Oxide, LPS and the Pathogenesis of Asthma - Phase II
Brief Title: Nitric Oxide, LPS and the Pathogenesis of Asthma Phase II
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding period completed.
Sponsor: John Sundy (Other)
Collaborators: Sandler Program for Asthma Research (Other)
Responsible Party: Sponsor-Investigator, John Sundy, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00005035; Pro00005035; 12496-CP-006B (Other: NIEHS)
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: LPS endotoxin
MeSH Terms: interventions — trinitrophenyl-lipopolysaccharide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Sterile Saline, LPS endotoxin
  Interventions: Biological: LPS endotoxin

INTERVENTIONS:
Biological: LPS endotoxin — Low challenge: saline (diluent), 5000EU, 10,000EU and 20,000EU LPS endotoxin as tolerated
  High challenge: Saline (diluent), 40,000EU and 80,000EU as tolerated
  Diluent Challenge: 3 X Sterile saline inhalation (2 ml)
  Other Names: Lipopolysaccaharide; Sterile Saline

SUMMARY:
The purpose of the study is to determine the role of nitric oxide (NO) in asthma and to characterize the symptoms associated with inhaled endotoxin (lipopolysaccharide [LPS]) in normal subjects. In this study, we will determine the effect of inhaled endotoxin on exhaled NO in healthy African Americans, with and without NOS2 promoter polymorphisms. The protocol described in this submission will involve the use of NIH Clinical Center Reference Endotoxin which has been approved by the FDA under IND BB-IND-10035.

DETAILED DESCRIPTION:
(IRB# Pro00005035)

The purpose of the study is to determine the role of nitric oxide (NO) in asthma and to characterize the symptoms associated with inhaled endotoxin in normal subjects. The effect of inhaled endotoxin on exhaled NO is determined in healthy African Americans, with and without NOS2 promoter polymorphisms. The protocol involves the use of NIH Clinical Center Reference Endotoxin which has been approved by the FDA under IND BB-IND-10035.

Background & significance: Asthma is a significant cause of morbidity and mortality for African Americans and asthma is increasing in prevalence. Both environmental and genetic factors contribute to the pathogenesis of asthma. In addition to allergens, environmental lipopolysaccharide (LPS) or endotoxin plays an important role in the chronic inflammation associated with asthma. There is convincing evidence that endotoxin exacerbates airflow obstruction and airway inflammation in allergic asthmatics. Endotoxin increases inducible nitric oxide synthase (NOS2) expression and nitric oxide (NO) production in vitro and in vivo in humans.

In asthma, NOS2 expression is upregulated in several cell types including bronchial epithelium, macrophages and other inflammatory cells. The increase in NOS2 expression is associated with increases in exhaled NO in individuals with asthma as compared to healthy individuals.

This prompted our search for NOS2 single nucleotide polymorphisms (SNPs) and the subsequent identification of three NOS2 promoter SNPs. Two of the SNPs are associated with increased systemic NO levels. Another SNP creates a predicted binding site for the human homolog of delta EF1, which is a transcriptional repressor and we predicted that this SNP would be associated with low NO levels. Importantly, the three NOS2 promoter SNPs are not linked, do not segregate together and are present primarily in individuals of African ancestry.

Design & procedures: The study of exhaled NO levels in individuals with asthma is confounded by the presence of cell types besides bronchial epithelium that produce NO, by differences in the severity of asthma and by the use of medications such as corticosteroids which alter exhaled NO levels. Therefore, in this protocol exhaled NO levels are measured in asymptomatic healthy African Americans.

Thirty individuals (10 individuals with each polymorphism) who are heterozygous for a NOS2 promoter SNPs and 10 individuals without these NOS2 promoter SNPs will be studied. The decision to study 10 individuals in each group was based on a power analysis (80% power, 0.05 alpha) using available data on NO levels in normal individuals following endotoxin challenge. Because basal NO levels in patients with asthma are approximately twice that of normal individuals, we decided that a two-fold difference in exhaled NO levels following endotoxin challenge represents a meaningful difference.

The general design of this study is to identify healthy nonasthmatic, nonatopic, never cigarette smokers with no history of airway reactivity, and subject them to a specific incremental challenge with inhaled LPS to determine the airway reactivity to inhaled endotoxin. Upon recruitment, each study subject will be scheduled for seven separate visits, with the option of 3 additional visits after each challenge. During the initial visit, each study participant will undergo a thorough clinical evaluation including 2 questionnaires, a physical examination, skin tests to assess the presence of atopy, full pulmonary function testing, a chest x-ray, an EKG, and a methacholine challenge test to assess airway hyperreactivity, exhaled nitric oxide and exhaled breath condensate samples to measure inflammatory mediators. During the challenge visits, each subject will undergo a specific incremental challenge with inhaled endotoxin or the vehicle (saline). The initial evaluation and the endotoxin inhalation challenge will be separated by a minimum of two weeks. A brief follow up visits will be scheduled to collect blood samples, exhaled gases 24, 48, 72hours and 7 days after endotoxin challenge and to obtain full pulmonary function testing with airway resistance performed at baseline. To avoid problems with diurnal variation in pulmonary function, all testing sessions will begin at 8:00 AM. All testing will be performed in the Rankin Duke Clinical Research Unit at Duke University. Serum pregnancy testing will be performed during the initial visit and the days of each endotoxin and saline inhalation challenge to exclude pregnant women from this study. Administration of endotoxin or saline will not occur until results of the pregnancy test have returned negative.

In addition to serum pregnancy testing, blood samples will be obtained to determine IgE levels (to determine whether subject has allergies; determined at visit 1 only), cotinine levels (a metabolite of nicotine and used to determine whether subject smokes; determined at visits 1, 2, 4 and 6), CRP and cytokine levels (markers of inflammation used to determine whether systemic responses to inhaled endotoxin occur; determined at visits 2, 3, 4, 5, 6 and 7), and RNA levels (to be analyzed using gene arrays and used to determine whether systemic responses to inhaled endotoxin occur; determined at visits 2, 3, 4, 5, 6 and 7). On visits 2, 4 and 6, CRP, cytokine and RNA levels will be determined three times, initially to establish baseline levels and 2 and 6 hours after endotoxin or saline challenge. On visits 3, 5 and 7, CRP, cytokine and RNA levels will be determined once. The URI questionnaire will be administered at the beginning of all visits to assess whether subjects have symptoms consistent with a URI or cold.

The Duke Investigational Pharmacy will prepare the inhaled solution of endotoxin according to a standard protocol which has been used successfully by other investigators, as well as in our own laboratory. Each subject will receive an initial dose of Saline Solution as a baseline. During the second visit, inhalations will contain increasing concentrations of endotoxin (Clinical Center Reference Endotoxin (CCRE), a lot of endotoxin prepared from the bacterial strain E. Coli O:113 and maintained by the Pharmaceutical Development Service, Warren Grant Magnuson Clinical Center, National Institutes of Health) according to the following schedule: 5,000 EU (endotoxin units); 10,000 EU; and 20,000 EU. During the higher dose challenge visit, inhalations will contain 40,000 EU and 80,000 EU of endotoxin. Following inhalation of each dose of endotoxin or each saline challenge, we will obtain several spirometric measures of airflow. Airflow will be assessed 1, 10, 20, and 30 minutes following each dose of inhaled LPS or saline. If the study subject's FEV1 is more than 80% of the baseline measurement, the inhalation challenge will continue and the next higher dose of endotoxin will be administered. During the control visit, saline control will be administered on three occasions. After each dose of inhaled endotoxin or saline, non-pulmonary adverse events will be assessed and graded. The protocol will conclude if any of the following criteria have been met: 1) subject does not wish to continue for any reason; 2) subject's FEV1 has decreased 20% from baseline saline inhalation; 3) total dose of 35,000 units (low dose challenge visit) or 120,000 units (high dose challenge visit) has been achieved; or 4) the subject experiences any adverse event rated as severe or any other adverse event deemed significant in the opinion of the investigator. Following completion of the inhaled endotoxin or saline challenge, pulmonary function studies, vital signs and symptom assessments will be performed to assess the safety of the inhaled endotoxin procedure (see attached IND protocol for details). We will also collect exhaled breath condensate samples to measure inflammatory mediators including leukotrienes and to control for the confounding effects of airway inflammation on exhaled NO levels. Exhaled breath condensate will be collected from subjects by having them breathe normally for approximately 10 minutes into an apparatus that traps condensation by cooling the exhaled breath. We will measure airway resistance at 1, 2, 6 and 24 hours after endotoxin or saline challenge. Measurement of spirometry, lung volumes, diffusing capacity will be repeated at 6 hours and 24 hours post challenge.

We will measure exhaled NO levels using an online chemiluminescent detector (Sievers 280i) prior to and 1, 2 and 6 hours after endotoxin or saline challenge. We will also measure exhaled NO levels 24 hours after exposure to endotoxin or saline.

Subjects will be requested to come for additional optional physiologic measurements at 48, 72 and 168 hours post challenge to gather data further in the time course. For the optional visits after each challenge, subjects will have vital signs measured, CRP and serum for other inflammatory markers drawn. Subjects will perform spirometry, lung volumes, diffusing capacity, exhaled NO levels, airway resistance, and complete a short questionnaire.

NOTE:

In a separate related IRB protocol prior to the above study:

In Phase 1, (IRB # Pro00005046) we will determine the effect of promoter polymorphisms in the gene for the NO producing enzyme, nitric oxide synthase (NOS2), on exhaled NO in healthy African Americans. Individuals consented during Phase 1 will be asked if they are willing to be contacted about future studies including those described in Phase 2 of this study. 30 individuals (10 individuals with each polymorphism) identified in Phase 1 who are heterozygous for a NOS2 promoter SNPs and 10 individuals without these NOS2 promoter SNPs will be studied.

Because SNPs in the TLR4 gene result in a lack of airway obstruction in response to endotoxin, we will genotype the 1000 DNA samples for the Asp299Gly and Thr399Ile TLR4 polymorphisms in Phase 1 and exclude these individuals from the studies proposed in Phase 2. Likewise, CD14 serves as a coreceptor for endotoxin and polymorphisms in the CD14 gene and promoter have been associated with asthma and responsiveness to endotoxin. Therefore, to control for this potential confounder in our analysis, we will also test whether polymorphisms in the CD14 gene and its promoter are associated with responsiveness to inhaled endotoxin.

ELIGIBILITY:
Inclusion Criteria:

* Willing/able to give informed consent & adhere to visit/protocol schedules
* non-atopic, non-asthmatic by PFT and allergy skin testing
* never cigarette smoker,
* no significant occupational exposure to respiratory irritants or toxins,
* no chronic illness
* no chronic use of medications (excluding contraceptive medication),
* no systemic corticosteroid use in the previous month,
* no historical or physical examination evidence of unstable cardiac or severe lung disease,
* Women of childbearing potential must have a negative serum pregnancy test
* baseline FEV1 > 80% of the predicted value,
* no clinically significant abnormalities on the chest x-ray or EKG

Exclusion Criteria:

* occupational exposure to hay or grain
* smoked 20 or more packs of cigarettes in a lifetime.
* prior allergen immunotherapy
* Allergy to potential study medications acetaminophen and albuterol
* Subjects who abuse alcohol or illicit substances will be excluded
* Viral respiratory infection within the previous 14 days
* Students or employees under direct supervision by protocol investigators are ineligible
* Nursing mothers
* Other investigational medication within the last 30 days
* Other medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2003-04; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Differential response to inhaled LPS based on NOS2 inhibition. | 24 hours with optional 48 hr,72hr and 7 day follow up

SECONDARY OUTCOMES:
Physiologic measurements | 24 hours with optional return up at 48 hrs, 72hrs and 7 day follow up

CONTACTS AND LOCATIONS:
Overall Officials: John C Sundy, M.D. PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States